CLINICAL TRIAL: NCT01369355
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Safety and Efficacy of Ustekinumab Maintenance Therapy in Subjects With Moderately to Severely Active Crohn's Disease
Brief Title: A Study to Evaluate the Safety and Efficacy of Ustekinumab Maintenance Therapy in Patients With Moderately to Severely Active Crohn's Disease (IM-UNITI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR018421; CNTO1275CRD3003 (Other: Janssen Research & Development, LLC); 2010-022760-12 (EudraCT Number)
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Crohn's Disease; Colitis; IBD; Inflammatory Bowel Disease
Keywords: Ustekinumab; Stelara, Moderately to severely active Crohn's Disease; IBD, Crohn's; UNITI; colitis; IL-12; IL-23
MeSH Terms: conditions — Crohn Disease; Colitis; Inflammatory Bowel Diseases | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (6):
- 001 (Placebo Comparator): Participants who were responders to Intravenous (IV) infusion of ustekinumab induction will be randomized to receive a single dose of placebo subcutaneously (SC) every 4 weeks (q4w).
  Interventions: Drug: Placebo SC
- 002 (Experimental): Participants who were responders to IV ustekinumab induction will be randomized to receive a single dose of ustekinumab 90 milligram (mg) SC every 12 weeks (q12w).
  Interventions: Drug: Ustekinumab 90 mg SC q12w
- 003 (Experimental): Participants who were responders to IV ustekinumab induction will be randomized to receive a single dose of ustekinumab 90 mg SC every 8 weeks (q8w).
  Interventions: Drug: Ustekinumab 90 mg SC q8w
- 004 (Experimental): Participants who were nonresponders to IV ustekinumab induction will receive a single dose of ustekinumab 90 mg SC and one placebo IV at week 0, if then respond will continue to receive one ustekinumab 90 mg SC q8w.
  Interventions: Drug: Placebo IV; Drug: Ustekinumab 90 mg SC q8w
- 005 (Experimental): Participants who were nonresponders to IV placebo induction will receive a single dose of ustekinumab 130 mg IV and one placebo SC at week 0, if then respond will continue to receive one ustekinumab 90 mg SC at week 8 then q12w.
  Interventions: Drug: Placebo SC; Drug: Ustekinumab 130 mg IV; Drug: Ustekinumab 90 mg SC q12w
- 006 (Placebo Comparator): Participants who were responders to IV placebo induction will receive one dose of placebo SC q4w.
  Interventions: Drug: Placebo SC

INTERVENTIONS:
Drug: Placebo SC — Placebo will be administered subcutaneously.
  Arms: 001; 005; 006
Drug: Placebo IV — Placebo will be administered as a single Intravenous infusion at week 0.
  Arms: 004
Drug: Ustekinumab 90 mg SC q8w — Ustekinumab 90 mg will be administered subcutaneously every 8 weeks (q8w) through Week 40.
  Arms: 003; 004
Drug: Ustekinumab 130 mg IV — Ustekinumab 130 mg will be administered as a single intravenous infusion at week 0.
  Arms: 005
Drug: Ustekinumab 90 mg SC q12w — Ustekinumab 90 mg will be administered as subcutaneously every 12 weeks (q12w) through Week 40.
  Arms: 002; 005

SUMMARY:
The primary purpose of this study is to evaluate the efficacy and safety of 2 maintenance regimens of ustekinumab administered subcutaneously to patients with moderately to severely active Crohn's disease who responded to treatment with intravenous ustekinumab in studies CNTO1275CRD3001 and CNTO1275CRD3002, compared to subcutaneously administered placebo.

DETAILED DESCRIPTION:
The main purpose of this study is to determine whether additional ustekinumab treatment is beneficial in patients with moderately to severely active Crohn's disease who initially had a clinical response to IV ustekinumab in one of the 2 initial induction studies (the CNTO1275CRD3001 ["UNITI-1"] or CNTO1275CRD3002 ["UNITI-2"] induction studies). The maintenance treatment will be injections in the skin (given subcutaneously, or "SC") of 90 mg ustekinumab either every 8 weeks or 12 weeks, and the effects (both the benefits and any side effects or adverse events) will be compared to SC placebo injections (otherwise identical except without ustekinumab). Patients who responded to IV ustekinumab in the UNITI-1 (NCT01369329) or UNITI-2 (NCT01369342) induction studies will be put into one of these 3 groups by chance (randomly, like rolling dice). The study will be double-blinded (so that neither patients nor study personnel know the identity of the assigned treatment). Patients who are randomized to either SC placebo or 90mg ustekinumab SC every 12 weeks who experience worsening in their Crohn's Disease symptoms (per the study loss of response criteria) will have their treatment adjusted so that they will instead start to receive 90mg ustekinumab SC every 8 weeks. All patients from the UNITI-1 or UNITI-2 studies (in addition to the patients described above who responded to IV ustekinumab) will be eligible to enter this study, provided the Week 8 visit in those trials was completed and study requirements are still met. Patients who are not in clinical response to IV placebo or ustekinumab in UNITI-1 or UNITI-2 will receive both IV and SC study agent at the first visit of this study (week 0). Patients previously receiving IV placebo will receive ustekinumab 130 mg IV at week 0 (and SC placebo), and patients previously receiving IV ustekinumab will receive 90 mg ustekinumab SC at week 0 (as well as IV placebo). If these patients are in clinical response 8 weeks later, they will receive 90 SC ustekinumab at that week8 visit, and will continue to receive Ustekinumab (every 8 weeks for participants not in response to IV Ustekinumab and every 12 weeks for participants not in response to IV Placebo) throughout the rest of the study (provided they otherwise remain eligible). Patients in clinical response to IV placebo induction dosing will continue to receive SC placebo. The main part of this study, also called the maintenance portion, will last 44 weeks. After week 44, all participants who are continuing to do well will be eligible to continue to receive study agent in the second part of the study, a long term extension where the study agent will continue to be administered up to week 252. Participants who discontinue study agent, either during the study, or after week 252, will be asked to return for a final safety follow-up visit 20 weeks after they last received study agent.

Patients in response to IV ustekinumab will be randomized to receive either placebo (Group 1), Ustekinumab 90 mg SC every 12 weeks (Group 2), or Ustekinumab 90mgSC every 8 weeks (Group 3). If patients in Groups 1 or 2 lose response, they will cross over to receive ustekinumab 90mg every 8 weeks. Other populations (nonresponders to prior IV ustekinumab or IV placebo) will receive ustekinumab at Week0 (either 90mg SC or 130mg IV, respectively) and continue SC ustekinumab if in response at Week 8, Placebo IV responders will continue to receive Placebo SC q4w.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received study agent at the start of study CNTO1275CRD3001 or CNTO1275CRD3002 and completed the Week 8 visit. Exclusion Criteria:
* Patients who underwent a Crohn's disease-related surgery since the start of induction study CNTO1275CRD3001 or CNTO1275CRD3002
* Patients who started a protocol prohibited medication since the start of studies CNTO1275CRD3001 and CNTO1275CRD3002
* Patients with protocol-specified changes to their concomitant medications due to Crohn's disease (due to lack of efficacy) since the start of studies CNTO1275CRD3001 and CNTO1275CRD3002

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1282 (Actual)
Dates: Start 2011-09-13 (Actual); Primary Completion 2015-06-10 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (220):
- United States (77):
  - Tucson, Arizona
  - La Jolla, California
  - Los Angeles, California
  - San Carlos, California
  - San Diego, California
  - Santa Monica, California
  - Lone Tree, Colorado
  - New Haven, Connecticut
  - Boca Raton, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Naples, Florida
  - Weston, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Macon, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Evanston, Illinois
  - Clive, Iowa
  - Pratt, Kansas
  - Crestview Hills, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Chevy Chase, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Chesterfield, Michigan
  - Detroit, Michigan
  - Troy, Michigan
  - Ypsilanti, Michigan
  - Rochester, Minnesota
  - Jackson, Mississippi
  - Ocean Springs, Mississippi
  - Columbia, Missouri
  - Lee's Summit, Missouri
  - Urbana, Missouri
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Marlton, New Jersey
  - Great Neck, New York
  - New York, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Mentor, Ohio
  - Oklahoma City, Oklahoma
  - Bend, Oregon
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - North Charleston, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - Grapevine, Texas
  - Houston, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Chesapeake, Virginia
  - Virginia Beach, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
- Australia (9):
  - Adelaide
  - Bedford Park
  - Box Hill
  - Central Queensland M C
  - Concord
  - Garran
  - Liverpool
  - Malvern
  - Parkville
- Austria (2):
  - Innsbruck
  - Vienna
- Belgium (3):
  - Brussels
  - Leuven
  - Liège
- Brazil (4):
  - Goiânia
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
- Bulgaria (4):
  - Pleven
  - Rousse
  - Sofia
  - Varna
- Canada (11):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Brandon, Manitoba
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Saskatoon, Saskatchewan
- Croatia (2):
  - Rijeka
  - Zagreb
- Czechia (2):
  - Hradec Králové
  - Ústí nad Labem
- Denmark (2):
  - Herlev
  - Silkeborg
- France (8):
  - Lille
  - Marseille
  - Paris
  - Pessac
  - Reims
  - Rouen
  - Toulouse
  - Vandœuvre-lès-Nancy
- Germany (18):
  - Berlin
  - Erlangen
  - Frankfurt
  - Freiburg im Breisgau
  - Halle
  - Hamburg
  - Hanover
  - Haßloch
  - Heidelberg
  - Jena
  - Kiel
  - LÿNEBURG
  - Mannheim
  - München
  - Münster
  - Regensburg
  - Stade
  - Ulm
- Hungary (7):
  - Békéscsaba
  - Budapest
  - Debrecen
  - Mosonmagyaróvár
  - Pécs
  - Szeksz Rd N/a
  - Székesfehérvár
- Reykjavik, Iceland
- Dublin, Ireland
- Israel (7):
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Tel Aviv
  - Tzrifin
- Japan (21):
  - Chikushino-shi
  - Fukuoka
  - Hachiōji
  - Hamamatsu
  - Hirosaki
  - Hiroshima
  - Kagoshima
  - Nishinomiya
  - Ohtsu
  - Osaka
  - Ōita
  - Sakura
  - Sapporo
  - Sendai
  - Suita-shi
  - Tokyo
  - Tsu
  - Uruma
  - Yokkaichi
  - Yokohama
  - Yokosuka
- Netherlands (3):
  - Amsterdam
  - Maastricht
  - Rotterdam
- New Zealand (7):
  - Auckland
  - Christchurch
  - Dunedin
  - Grafton
  - Hamilton
  - Hastings
  - Plenty
- Poland (4):
  - Elblag
  - Krakow
  - Lodz
  - Warsaw
- Russia (3):
  - Moscow
  - Novosibirsk
  - Saint Petersburg
- Belgrade, Serbia
- South Africa (4):
  - Cape Town
  - Cape Town Western Cape
  - Pretoria
  - Somerset West
- South Korea (3):
  - Daegu
  - Gyeonggi-do
  - Seoul
- Madrid, Spain
- United Kingdom (15):
  - Birmingham
  - Brighton
  - Bristol
  - Cambridge
  - Cardiff
  - Exeter
  - Gloucester
  - Liverpool
  - London
  - Manchester
  - Norwich
  - Nottinghamshirecc
  - Oxford
  - Shropshire
  - Southampton

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Timmer A. Anti-IL-12/23p40 antibodies for induction of remission in Crohn's disease. Cochrane Database Syst Rev. 2025 May 13;5(5):CD007572. doi: 10.1002/14651858.CD007572.pub4. PMID 40357993
- [Derived] Ghosh S, Feagan BG, Ott E, Gasink C, Godwin B, Marano C, Miao Y, Ma T, Loftus EV Jr, Sandborn WJ, Danese S, Abreu MT, Sands BE. Safety of Ustekinumab in Inflammatory Bowel Disease: Pooled Safety Analysis Through 5 Years in Crohn's Disease and 4 Years in Ulcerative Colitis. J Crohns Colitis. 2024 Aug 6;18(7):1091-1101. doi: 10.1093/ecco-jcc/jjae013. PMID 38310565
- [Derived] Colombel JF, Sands BE, Gasink C, Yeager B, Adedokun OJ, Izanec J, Ma T, Gao LL, Lee SD, Targan SR, Ghosh S, Hanauer SB, Sandborn WJ. Evolution of Symptoms After Ustekinumab Induction Therapy in Patients With Crohn's Disease. Clin Gastroenterol Hepatol. 2024 Jan;22(1):144-153.e2. doi: 10.1016/j.cgh.2023.06.014. Epub 2023 Jun 28. PMID 37391056
- [Derived] Dubinsky M, Ma C, Griffith J, Crowell M, Neimark E, Kligys K, O'Connell T. Matching-Adjusted Indirect Comparison Between Risankizumab and Ustekinumab for Induction and Maintenance Treatment of Moderately to Severely Active Crohn's Disease. Adv Ther. 2023 Sep;40(9):3896-3911. doi: 10.1007/s12325-023-02546-6. Epub 2023 Jun 27. PMID 37368103
- [Derived] Adedokun OJ, Xu Z, Gasink C, Kowalski K, Sandborn WJ, Feagan B. Population Pharmacokinetics and Exposure-Response Analyses of Ustekinumab in Patients With Moderately to Severely Active Crohn's Disease. Clin Ther. 2022 Oct;44(10):1336-1355. doi: 10.1016/j.clinthera.2022.08.010. Epub 2022 Sep 21. PMID 36150926
- [Derived] Narula N, Aruljothy A, Wong ECL, Homenauth R, Alshahrani AA, Marshall JK, Reinisch W. The impact of ustekinumab on extraintestinal manifestations of Crohn's disease: A post hoc analysis of the UNITI studies. United European Gastroenterol J. 2021 Jun;9(5):581-589. doi: 10.1002/ueg2.12094. Epub 2021 Jun 2. PMID 34077627
- [Derived] Sandborn WJ, Rebuck R, Wang Y, Zou B, Adedokun OJ, Gasink C, Sands BE, Hanauer SB, Targan S, Ghosh S, de Villiers WJS, Colombel JF, Feagan BG, Lynch JP. Five-Year Efficacy and Safety of Ustekinumab Treatment in Crohn's Disease: The IM-UNITI Trial. Clin Gastroenterol Hepatol. 2022 Mar;20(3):578-590.e4. doi: 10.1016/j.cgh.2021.02.025. Epub 2021 Feb 19. PMID 33618023
- [Derived] Sandborn WJ, Feagan BG, Danese S, O'Brien CD, Ott E, Marano C, Baker T, Zhou Y, Volger S, Tikhonov I, Gasink C, Sands BE, Ghosh S. Safety of Ustekinumab in Inflammatory Bowel Disease: Pooled Safety Analysis of Results from Phase 2/3 Studies. Inflamm Bowel Dis. 2021 Jun 15;27(7):994-1007. doi: 10.1093/ibd/izaa236. PMID 32964215
- [Derived] Li K, Friedman JR, Chan D, Pollack P, Yang F, Jacobstein D, Brodmerkel C, Gasink C, Feagan BG, Sandborn WJ, Rutgeerts P, De Hertogh G. Effects of Ustekinumab on Histologic Disease Activity in Patients With Crohn's Disease. Gastroenterology. 2019 Oct;157(4):1019-1031.e7. doi: 10.1053/j.gastro.2019.06.037. Epub 2019 Jul 4. PMID 31279870
- [Derived] Hanauer SB, Sandborn WJ, Feagan BG, Gasink C, Jacobstein D, Zou B, Johanns J, Adedokun OJ, Sands BE, Rutgeerts P, de Villiers WJS, Colombel JF, Ghosh S. IM-UNITI: Three-year Efficacy, Safety, and Immunogenicity of Ustekinumab Treatment of Crohn's Disease. J Crohns Colitis. 2020 Jan 1;14(1):23-32. doi: 10.1093/ecco-jcc/jjz110. PMID 31158271
- [Derived] Ghosh S, Gensler LS, Yang Z, Gasink C, Chakravarty SD, Farahi K, Ramachandran P, Ott E, Strober BE. Ustekinumab Safety in Psoriasis, Psoriatic Arthritis, and Crohn's Disease: An Integrated Analysis of Phase II/III Clinical Development Programs. Drug Saf. 2019 Jun;42(6):751-768. doi: 10.1007/s40264-019-00797-3. PMID 30739254
- [Derived] Rutgeerts P, Gasink C, Chan D, Lang Y, Pollack P, Colombel JF, Wolf DC, Jacobstein D, Johanns J, Szapary P, Adedokun OJ, Feagan BG, Sandborn WJ. Efficacy of Ustekinumab for Inducing Endoscopic Healing in Patients With Crohn's Disease. Gastroenterology. 2018 Oct;155(4):1045-1058. doi: 10.1053/j.gastro.2018.06.035. Epub 2018 Aug 29. PMID 29909019
- [Derived] Sandborn WJ, Rutgeerts P, Gasink C, Jacobstein D, Zou B, Johanns J, Sands BE, Hanauer SB, Targan S, Ghosh S, de Villiers WJS, Colombel JF, Feagan BG. Long-term efficacy and safety of ustekinumab for Crohn's disease through the second year of therapy. Aliment Pharmacol Ther. 2018 Jul;48(1):65-77. doi: 10.1111/apt.14794. Epub 2018 May 24. PMID 29797519
- [Derived] Adedokun OJ, Xu Z, Gasink C, Jacobstein D, Szapary P, Johanns J, Gao LL, Davis HM, Hanauer SB, Feagan BG, Ghosh S, Sandborn WJ. Pharmacokinetics and Exposure Response Relationships of Ustekinumab in Patients With Crohn's Disease. Gastroenterology. 2018 May;154(6):1660-1671. doi: 10.1053/j.gastro.2018.01.043. Epub 2018 Feb 1. PMID 29409871
- [Derived] Hibi T, Imai Y, Murata Y, Matsushima N, Zheng R, Gasink C. Efficacy and safety of ustekinumab in Japanese patients with moderately to severely active Crohn's disease: a subpopulation analysis of phase 3 induction and maintenance studies. Intest Res. 2017 Oct;15(4):475-486. doi: 10.5217/ir.2017.15.4.475. Epub 2017 Oct 23. PMID 29142515
- [Derived] Feagan BG, Sandborn WJ, Gasink C, Jacobstein D, Lang Y, Friedman JR, Blank MA, Johanns J, Gao LL, Miao Y, Adedokun OJ, Sands BE, Hanauer SB, Vermeire S, Targan S, Ghosh S, de Villiers WJ, Colombel JF, Tulassay Z, Seidler U, Salzberg BA, Desreumaux P, Lee SD, Loftus EV Jr, Dieleman LA, Katz S, Rutgeerts P; UNITI-IM-UNITI Study Group. Ustekinumab as Induction and Maintenance Therapy for Crohn's Disease. N Engl J Med. 2016 Nov 17;375(20):1946-1960. doi: 10.1056/NEJMoa1602773. PMID 27959607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 1282 participants enrolled,1 was excluded from study before assignment to arm/group due to deviation from Good Clinical Practice at 1 study site. Hence 1281 participants were analyzed. Total 397 participants who were in clinical response to ustekinumab induction were randomized in maintenance study and considered as primary population.
Pre-assignment Details: Due to a stability issue with the batch of Intravenous (IV) drug (130 mg ustekinumab), in November 2011 sponsor temporarily suspended dosing in induction studies (CRD3001 and CRD3002) and this maintenance study (CRD3003). All 3 studies were restarted with a 90 milligram per milliliter (mg/mL) formulation for IV administration on 17 February 2012.
Groups:
- Ustekinumab Induction Responders(UST-I-Rsp)Placebo Maintenance: Participants (who were in clinical response to ustekinumab IV at Week 8 of an induction study) randomized to receive placebo subcutaneously (SC) every 4 weeks (q4w) in the maintenance study.
- UST-I-Rsp-UST-90 mg Every 12 Weeks (Q12W) Maintenance: Participants (who were in clinical response to ustekinumab IV at Week 8 of an induction study) randomized to receive ustekinumab SC 90 milligrams (mg) q12w in the maintenance study.
- UST-I-Rsp-UST-90 mg Q8W Maintenance: Participants (who were in clinical response to ustekinumab IV at Week 8 of an induction study) randomized to receive ustekinumab SC 90 mg q8w in the maintenance study.
- Placebo (PBO)-I-Rsp - PBO Maintenance: Participants (who were in clinical response to placebo IV at Week 8 of an induction study) received placebo SC q4w in the maintenance study; not randomized.
- PBO-I-nonRsp - UST-130mg Intravenous/90mg SC Q12W Maintenance: Participants (who were not in clinical response to placebo IV at Week 8 of an induction study) received ustekinumab 130 mg IV on entry into maintenance followed by ustekinumab 90 mg SC q12 weeks beginning at Week 8 of maintenance (if in response); not randomized.
- UST-I-nonRsp - UST-90mg Subcutaneously (SC) Q8W Maintenance: Participants (who were not in clinical response to ustekinumab IV at Week 8 of an induction study) received ustekinumab 90 mg SC on entry into maintenance followed by ustekinumab 90 mg SC q8w beginning at Week 8 of maintenance (if in response); not randomized.
- Placebo Long Term Extension (LTE): Participants who received placebo SC in the maintenance study, entered the LTE and continued to receive placebo SC in the LTE study (Week 44 to 272).
- UST 90 mg SC Q12W LTE: Participants entered the LTE and continued to receive ustekinumab 90 mg SC q12w in the LTE study (Week 44 to 272).
- UST 90 mg SC Q8W LTE: Participants entered the LTE and continued to receive ustekinumab 90 mg SC q8w in the LTE study (Week 44 to 272).
Period: Week 0 - Week 44 (Maintenance)
Arm/Group | Ustekinumab Induction Responders(UST-I-Rsp)Placebo Maintenance | UST-I-Rsp-UST-90 mg Every 12 Weeks (Q12W) Maintenance | UST-I-Rsp-UST-90 mg Q8W Maintenance | Placebo (PBO)-I-Rsp - PBO Maintenance | PBO-I-nonRsp - UST-130mg Intravenous/90mg SC Q12W Maintenance | UST-I-nonRsp - UST-90mg Subcutaneously (SC) Q8W Maintenance | Placebo Long Term Extension (LTE) | UST 90 mg SC Q12W LTE | UST 90 mg SC Q8W LTE
Started | 133 | 132 | 132 | 123 | 285 | 476 | 0 | 0 | 0
Completed | 102 | 103 | 101 | 93 | 131 | 204 | 0 | 0 | 0
Not Completed | 31 | 29 | 31 | 30 | 154 | 272 | 0 | 0 | 0
Not completed — Adverse Event | 9 | 12 | 6 | 7 | 14 | 25 | 0 | 0 | 0
Not completed — Lack of Efficacy | 15 | 14 | 15 | 15 | 126 | 217 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 2 | 5 | 6 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 7 | 6 | 8 | 22 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Period: Long-term Extension (Week 44-272)
Arm/Group | Ustekinumab Induction Responders(UST-I-Rsp)Placebo Maintenance | UST-I-Rsp-UST-90 mg Every 12 Weeks (Q12W) Maintenance | UST-I-Rsp-UST-90 mg Q8W Maintenance | Placebo (PBO)-I-Rsp - PBO Maintenance | PBO-I-nonRsp - UST-130mg Intravenous/90mg SC Q12W Maintenance | UST-I-nonRsp - UST-90mg Subcutaneously (SC) Q8W Maintenance | Placebo Long Term Extension (LTE) | UST 90 mg SC Q12W LTE | UST 90 mg SC Q8W LTE
Started | 0 | 0 | 0 | 0 | 0 | 0 | 151 | 213 | 354
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 107 | 183
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 151 | 106 | 171
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 29 | 53
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 26 | 29
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 11
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 30 | 47
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 110 | 9 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ustekinumab Induction Responders(UST-I-Rsp)Placebo Maintenance | UST-I-Rsp-UST-90 mg Every 12 Weeks (Q12W) Maintenance | UST-I-Rsp-UST-90 mg Q8W Maintenance | Placebo (PBO)-I-Rsp - PBO Maintenance | PBO-I-nonRsp - UST-130mg Intravenous/90mg SC Q12W Maintenance | UST-I-nonRsp - UST-90mg Subcutaneously (SC) Q8W Maintenance | Total
Number analyzed (Participants) | 133 | 132 | 132 | 123 | 285 | 476 | 1281
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (12.69) | 38.6 (13.65) | 37.9 (13.2) | 39.1 (12.46) | 39 (12.33) | 37.4 (12.5) | 38.3 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 74 | 76 | 64 | 149 | 275 | 712
  Male | 59 | 58 | 56 | 59 | 136 | 201 | 569
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 4 | 2 | 3 | 4 | 10 | 15 | 38
  Austria | 1 | 3 | 1 | 0 | 0 | 1 | 6
  Belgium | 2 | 4 | 1 | 1 | 7 | 16 | 31
  Bulgaria | 5 | 2 | 2 | 4 | 1 | 7 | 21
  Brazil | 1 | 1 | 3 | 2 | 2 | 3 | 12
  Canada | 10 | 4 | 12 | 5 | 17 | 44 | 92
  Denmark | 1 | 2 | 1 | 0 | 0 | 0 | 4
  Spain | 1 | 0 | 1 | 0 | 0 | 1 | 3
  France | 6 | 8 | 9 | 1 | 13 | 27 | 64
  United Kingdom | 4 | 7 | 5 | 7 | 15 | 29 | 67
  Croatia | 1 | 1 | 0 | 1 | 0 | 1 | 4
  Hungary | 11 | 8 | 8 | 10 | 14 | 13 | 64
  Ireland | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Iceland | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Israel | 3 | 1 | 0 | 1 | 2 | 8 | 15
  Italy | 6 | 2 | 2 | 1 | 4 | 8 | 23
  Japan | 4 | 8 | 9 | 4 | 18 | 31 | 74
  Korea, Democratic People'S Republic Of | 3 | 3 | 2 | 2 | 5 | 7 | 22
  Netherlands | 4 | 4 | 4 | 1 | 9 | 14 | 36
  New Zealand | 3 | 5 | 2 | 1 | 1 | 3 | 15
  Poland | 3 | 5 | 6 | 6 | 6 | 10 | 36
  Russia | 2 | 2 | 3 | 5 | 1 | 4 | 17
  Serbia | 2 | 7 | 4 | 3 | 2 | 1 | 19
  United States | 41 | 42 | 40 | 50 | 124 | 198 | 495
  South Africa | 5 | 2 | 5 | 7 | 5 | 7 | 31
  Czech Republic | 0 | 0 | 1 | 0 | 2 | 2 | 5
  Germany | 9 | 8 | 7 | 7 | 27 | 26 | 84

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Remission at Week 44
Description: Clinical remission at Week 44 was defined as a Crohn's Disease Activity Index (CDAI) score of <150 points (in general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities). CDAI was assessed by collecting information on 8 different Crohn's disease-related variables (extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being). A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Week 44
Population: The primary efficacy analysis population in this study was randomized participants (i.e., participants who were in clinical response to ustekinumab induction dosing at Week 8 from one of the induction studies CRD3001 and CRD3002) after study restart.
Measure: Number; unit: participants
Groups:
- Placebo Subcutaneously (SC): Participants (who were in clinical response to ustekinumab IV at Week 8 of an induction study) randomized to receive placebo subcutaneously (SC) every 4 weeks (q4w) in the maintenance study.
- Ustekinumab 90 Milligram (mg) SC Every 12 Weeks (q12w): Participants (who were in clinical response to ustekinumab IV at Week 8 of an induction study) randomized to receive ustekinumab SC 90 mg q12w in the maintenance study.
- Ustekinumab 90 mg SC q8w: Participants (who were in clinical response to ustekinumab IV at Week 8 of an induction study) randomized to receive ustekinumab SC 90 mg q8w in the maintenance study.
Arm/Group | Placebo Subcutaneously (SC) | Ustekinumab 90 Milligram (mg) SC Every 12 Weeks (q12w) | Ustekinumab 90 mg SC q8w
Number analyzed (Participants) | 131 | 129 | 128
participants | 47 | 63 | 68
Statistical Analysis 1: Comparison: Placebo Subcutaneously (SC) vs Ustekinumab 90 Milligram (mg) SC Every 12 Weeks (q12w); Test type: Superiority or Other; p = 0.040, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; 2-sided Cochran-Mantel-Haenszel chi-square test, stratified by clinical remission at Week 0, ustekinumab induction dose and the induction study
Statistical Analysis 2: Comparison: Placebo Subcutaneously (SC) vs Ustekinumab 90 mg SC q8w; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants With Clinical Response at Week 44
Description: Clinical response at Week 44 was defined as a reduction from baseline in the Crohn's Disease Activity Index (CDAI) score of greater than or equal (>=) 100 points. Participants with a baseline CDAI score of > = 220 to less than or equal (< =) 248 were considered to be in clinical response if a CDAI score of less than (<) 150 was attained. A CDAI score of less than 150 indicates clinical remission. A decrease in CDAI score over time indicates improvement in disease activity.
Time Frame: Week 44
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo Subcutaneously (SC) | Ustekinumab 90 Milligram (mg) SC Every 12 Weeks (q12w) | Ustekinumab 90 mg SC q8w
Number analyzed (Participants) | 131 | 129 | 128
participants | 58 | 75 | 76
Statistical Analysis 1: Comparison: Placebo Subcutaneously (SC) vs Ustekinumab 90 Milligram (mg) SC Every 12 Weeks (q12w); Test type: Superiority or Other; p = 0.033, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo Subcutaneously (SC) vs Ustekinumab 90 mg SC q8w; Test type: Superiority or Other; p = 0.018, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants in Clinical Remission at Week 44 Among Participants in Clinical Remission to Ustekinumab at Week 0 of Maintenance Study
Description: Clinical remission at week 44 was defined as a CDAI score of < 150 points among participants in clinical remission to ustekinumab at week 0 of maintenance study.
Time Frame: Week 44
Population: Analysis population included all randomized participants after the study was restarted (who were in clinical remission at Week 0 of maintenance study). 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Placebo Subcutaneously (SC) | Ustekinumab 90 Milligram (mg) SC Every 12 Weeks (q12w) | Ustekinumab 90 mg SC q8w
Number analyzed (Participants) | 79 | 78 | 78
participants | 36 | 44 | 52
Statistical Analysis 1: Comparison: Placebo Subcutaneously (SC) vs Ustekinumab 90 Milligram (mg) SC Every 12 Weeks (q12w); Test type: Superiority or Other; p = 0.189, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; 2-sided Cochran-Mantel-Haenszel chi-square test, stratified by ustekinumab induction dose and the induction study
Statistical Analysis 2: Comparison: Placebo Subcutaneously (SC) vs Ustekinumab 90 mg SC q8w; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; 2-sided Cochran-Mantel-Haenszel chi-square test, stratified by ustekinumab induction dose and the induction study

4. Secondary Outcome: Number of Participants With Corticosteroid-free Remission at Week 44
Description: Corticosteroid-free remission at Week 44 was defined as a CDAI score of <150 points without receiving corticosteroids at Week 44.
Time Frame: Week 44
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo Subcutaneously (SC) | Ustekinumab 90 Milligram (mg) SC Every 12 Weeks (q12w) | Ustekinumab 90 mg SC q8w
Number analyzed (Participants) | 131 | 129 | 128
participants | 39 | 55 | 60
Statistical Analysis 1: Comparison: Placebo Subcutaneously (SC) vs Ustekinumab 90 Milligram (mg) SC Every 12 Weeks (q12w); Test type: Superiority or Other; p = 0.035, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo Subcutaneously (SC) vs Ustekinumab 90 mg SC q8w; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants in Clinical Remission at Week 44 in the Subset of Participants Who Were Refractory or Intolerant to Tumor Necrosis Factor (TNF) Antagonist Therapy
Description: Clinical remission at Week 44 was defined as a CDAI score of <150 points in the subset of participants who were refractory or Intolerant to tumor necrosis factor antagonist therapy.
Time Frame: Week 44
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo Subcutaneously (SC) | Ustekinumab 90 Milligram (mg) SC Every 12 Weeks (q12w) | Ustekinumab 90 mg SC q8w
Number analyzed (Participants) | 61 | 57 | 56
participants | 16 | 22 | 23
Statistical Analysis 1: Comparison: Placebo Subcutaneously (SC) vs Ustekinumab 90 Milligram (mg) SC Every 12 Weeks (q12w); Test type: Superiority or Other; p = 0.140, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; 2 sided Cochran-Mantel-Haenszel chi-square test, stratified by clinical remission status at Week 0 and ustekinumab induction dose
Statistical Analysis 2: Comparison: Placebo Subcutaneously (SC) vs Ustekinumab 90 mg SC q8w; Test type: Superiority or Other; p = 0.102, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to Week 272
Description: Safety was analyzed for all treated participants who received at least 1 administration of study agent in the maintenance (Week 0-44) and LTE study (Week 44-272).
Groups:
- Ustekinumab Induction Responders(USTIRsp) Placebo Maintenance: Participants (who were in clinical response to ustekinumab IV at Week 8 of an induction study) received placebo subcutaneously (SC) every 4 weeks (q4w) in the maintenance study (includes events up to the time of loss of response).
- UST -I-Rsp -PBO Maintenance -UST-90mg SC Q8W- Maintenance: Participants (who were in clinical response to ustekinumab IV at Week 8 of an induction study) received placebo SC and had dose adjustment to ustekinumab SC 90 mg q8w (includes events from the time of loss of response onward).
- UST-I-Rsp-UST 90 mg SC Every 12 Weeks (Q12W) Maintenance: Participants (who were in clinical response to ustekinumab IV at Week 8 of an induction study) received ustekinumab SC 90 milligrams (mg) q12w in the maintenance study (includes events up to the time of loss of response).
- UST-I-Rsp-UST 90 mg SC Q12W/Q8W Maintenance: Participants (who were in clinical response to ustekinumab IV at Week 8 of an induction study) received ustekinumab SC 90 mg q12w and had dose adjustment to ustekinumab SC 90 mg q8w in the maintenance study (includes events from the time of loss of response onward).
- UST-I-Rsp-UST 90 mg SC Q8W Maintenance: Participants (who were in clinical response to ustekinumab IV at Week 8 of an induction study) received ustekinumab SC 90 mg q8w (includes events up to the time of loss of response).
- UST IV-I-Rsp-UST-90mg Maintenance-UST-90mg SC Q8W Maintenance: Participants (who were in clinical response to ustekinumab IV at Week 8 of an induction study) received ustekinumab SC 90 mg q8 weeks and remained on ustekinumab 90 mg q8w upon loss of response (includes events from the time of loss of response onward).
- Placebo (PBO)-I-Rsp PBO Maintenance: Participants (who were in clinical response to placebo IV at Week 8 of an induction study) received placebo SC; not randomized.
- PBO-I-nonRsp- UST-130mg Intravenous/90mg SC Q12W Maintenance: Participants (who were not in clinical response to placebo IV at Week 8 of an induction study) received ustekinumab 130 mg IV on entry into maintenance followed by ustekinumab 90 mg SC q12 weeks beginning at Week 8 of maintenance (if in response); not randomized.
- UST IV-I-nonRsp - UST-90 mg SC Q8W Maintenance: Participants (who were not in clinical response to ustekinumab IV at Week 8 of an induction study) received ustekinumab 90 mg SC on entry into maintenance followed by ustekinumab 90 mg SC q8w beginning at Week 8 of maintenance (if in response); not randomized.
Arm/Group | Ustekinumab Induction Responders(USTIRsp) Placebo Maintenance | UST -I-Rsp -PBO Maintenance -UST-90mg SC Q8W- Maintenance | UST-I-Rsp-UST 90 mg SC Every 12 Weeks (Q12W) Maintenance | UST-I-Rsp-UST 90 mg SC Q12W/Q8W Maintenance | UST-I-Rsp-UST 90 mg SC Q8W Maintenance | UST IV-I-Rsp-UST-90mg Maintenance-UST-90mg SC Q8W Maintenance | Placebo (PBO)-I-Rsp PBO Maintenance | PBO-I-nonRsp- UST-130mg Intravenous/90mg SC Q12W Maintenance | UST IV-I-nonRsp - UST-90 mg SC Q8W Maintenance | Placebo Long Term Extension (LTE) | UST 90 mg SC Q12W LTE | UST 90 mg SC Q8W LTE
All-Cause Mortality (participants affected / at risk) | 0/133 | 0/51 | 0/132 | 0/29 | 0/131 | 0/29 | 0/123 | 0/285 | 0/476 | 0/151 | 2/213 | 4/354
Serious Adverse Events (participants affected / at risk) | 22/133 | 7/51 | 16/132 | 5/29 | 13/131 | 6/29 | 19/123 | 47/285 | 77/476 | 26/151 | 68/213 | 99/354
Other Adverse Events (participants affected / at risk) | 94/133 | 34/51 | 88/132 | 20/29 | 84/131 | 18/29 | 82/123 | 160/285 | 275/476 | 83/151 | 162/213 | 293/354
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ustekinumab Induction Responders(USTIRsp) Placebo Maintenance (N=133) | UST -I-Rsp -PBO Maintenance -UST-90mg SC Q8W- Maintenance (N=51) | UST-I-Rsp-UST 90 mg SC Every 12 Weeks (Q12W) Maintenance (N=132) | UST-I-Rsp-UST 90 mg SC Q12W/Q8W Maintenance (N=29) | UST-I-Rsp-UST 90 mg SC Q8W Maintenance (N=131) | UST IV-I-Rsp-UST-90mg Maintenance-UST-90mg SC Q8W Maintenance (N=29) | Placebo (PBO)-I-Rsp PBO Maintenance (N=123) | PBO-I-nonRsp- UST-130mg Intravenous/90mg SC Q12W Maintenance (N=285) | UST IV-I-nonRsp - UST-90 mg SC Q8W Maintenance (N=476) | Placebo Long Term Extension (LTE) (N=151) | UST 90 mg SC Q12W LTE (N=213) | UST 90 mg SC Q8W LTE (N=354)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aortic Valve Incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fibrous Dysplasia of Bone (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chorioretinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal Detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Strabismus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 5
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal Fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal Fistula (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colon Dysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Crohn's Disease (Gastrointestinal disorders) | 7 | 4 | 5 | 3 | 4 | 3 | 6 | 15 | 30 | 12 | 17 | 32
Cyclic Vomiting Syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterocutaneous Fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterovesical Fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epiploic Appendagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Fistula of Small Intestine (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ileal Stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Inflammatory Bowel Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal Stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Large Intestinal Stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal Stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal Prolapse (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal Stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 10 | 4 | 6 | 10
Small Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small Intestinal Stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Tooth Impacted (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysplasia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Incarcerated Hernia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Sudden Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bile Duct Stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1
Abdominal Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess Intestinal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal Abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 6 | 3
Anal Fistula Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Campylobacter Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Clostridium Difficile Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytomegalovirus Colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cytomegalovirus Viraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hepatitis Infectious Mononucleosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mastitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myringitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ophthalmic Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parainfluenzae Virus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Perirectal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 2
Pneumonia Pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia Staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Postoperative Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomembranous Colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rectal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Septic Shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tubo-Ovarian Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular Device Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Allergic Transfusion Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anastomotic Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anastomotic Leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal Anastomotic Stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Heat Stroke (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal Anastomosis Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural Intestinal Perforation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sternal Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Electrolytes Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Faecal Volume Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Troponin Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral Disc Space Narrowing (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign Neoplasm of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fibroadenoma of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lentigo Maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small Intestine Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dementia with Lewy Bodies (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Idiopathic Intracranial Hypertension (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intracranial Aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Trigeminal Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Premature Delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Premature Labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
End Stage Renal Disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1
Renal Colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal Tubular Necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bartholin's Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic Congestion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pulmonary Granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary Haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pustular Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast Prosthesis User (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Miscarriage of Partner (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Substance Abuser (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Hernia Repair (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileostomy Closure (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Knee Arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic Pouch Procedure (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rotator Cuff Repair (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aortic Dissection (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aortic Stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2
Essential Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypertensive Urgency (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ustekinumab Induction Responders(USTIRsp) Placebo Maintenance (N=133) | UST -I-Rsp -PBO Maintenance -UST-90mg SC Q8W- Maintenance (N=51) | UST-I-Rsp-UST 90 mg SC Every 12 Weeks (Q12W) Maintenance (N=132) | UST-I-Rsp-UST 90 mg SC Q12W/Q8W Maintenance (N=29) | UST-I-Rsp-UST 90 mg SC Q8W Maintenance (N=131) | UST IV-I-Rsp-UST-90mg Maintenance-UST-90mg SC Q8W Maintenance (N=29) | Placebo (PBO)-I-Rsp PBO Maintenance (N=123) | PBO-I-nonRsp- UST-130mg Intravenous/90mg SC Q12W Maintenance (N=285) | UST IV-I-nonRsp - UST-90 mg SC Q8W Maintenance (N=476) | Placebo Long Term Extension (LTE) (N=151) | UST 90 mg SC Q12W LTE (N=213) | UST 90 mg SC Q8W LTE (N=354)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 5 | 1 | 3 | 0 | 5 | 6 | 11 | 2 | 15 | 17
Abdominal Pain (Gastrointestinal disorders) | 17 | 3 | 12 | 5 | 11 | 1 | 15 | 23 | 38 | 16 | 38 | 68
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 1 | 4 | 1 | 2 | 2 | 5 | 8 | 15 | 8 | 11 | 22
Constipation (Gastrointestinal disorders) | 4 | 1 | 6 | 2 | 3 | 0 | 0 | 6 | 10 | 0 | 9 | 22
Crohn's Disease (Gastrointestinal disorders) | 12 | 5 | 12 | 3 | 12 | 2 | 13 | 17 | 40 | 25 | 44 | 80
Diarrhoea (Gastrointestinal disorders) | 7 | 2 | 11 | 1 | 5 | 0 | 11 | 10 | 12 | 11 | 30 | 50
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 1 | 0 | 2 | 4 | 7 | 2 | 11 | 15
Nausea (Gastrointestinal disorders) | 9 | 3 | 10 | 3 | 4 | 1 | 12 | 15 | 46 | 12 | 23 | 34
Vomiting (Gastrointestinal disorders) | 9 | 3 | 5 | 2 | 4 | 2 | 5 | 6 | 33 | 2 | 14 | 26
Fatigue (General disorders) | 6 | 2 | 8 | 1 | 6 | 0 | 9 | 11 | 15 | 8 | 13 | 29
Injection Site Erythema (General disorders) | 0 | 1 | 1 | 1 | 7 | 1 | 2 | 5 | 7 | 1 | 7 | 7
Pyrexia (General disorders) | 11 | 2 | 11 | 3 | 9 | 1 | 12 | 16 | 25 | 9 | 19 | 19
Bronchitis (Infections and infestations) | 4 | 3 | 1 | 0 | 6 | 0 | 3 | 5 | 7 | 4 | 13 | 30
Gastroenteritis (Infections and infestations) | 5 | 1 | 3 | 0 | 4 | 0 | 4 | 8 | 18 | 7 | 21 | 41
Gastroenteritis Viral (Infections and infestations) | 1 | 3 | 4 | 0 | 4 | 2 | 5 | 6 | 6 | 2 | 11 | 12
Influenza (Infections and infestations) | 4 | 1 | 8 | 1 | 5 | 1 | 4 | 9 | 8 | 4 | 25 | 37
Nasopharyngitis (Infections and infestations) | 10 | 4 | 17 | 4 | 14 | 0 | 15 | 32 | 52 | 16 | 54 | 100
Pharyngitis Streptococcal (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 2 | 2 | 3 | 1 | 0 | 2 | 3
Sinusitis (Infections and infestations) | 2 | 0 | 6 | 2 | 4 | 2 | 5 | 12 | 17 | 8 | 19 | 36
Upper Respiratory Tract Infection (Infections and infestations) | 21 | 1 | 9 | 0 | 13 | 1 | 7 | 25 | 33 | 14 | 40 | 62
Urinary Tract Infection (Infections and infestations) | 3 | 1 | 9 | 1 | 4 | 1 | 7 | 5 | 17 | 7 | 15 | 35
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 2 | 1 | 0 | 2 | 1 | 5 | 5 | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 6 | 22 | 5 | 18 | 3 | 23 | 29 | 49 | 11 | 27 | 40
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3 | 0 | 1 | 0 | 8 | 7 | 3 | 1 | 1 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 5 | 1 | 6 | 3 | 2 | 12 | 15 | 13 | 18 | 48
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 5 | 1 | 0 | 4 | 6 | 1 | 9 | 18
Headache (Nervous system disorders) | 15 | 6 | 15 | 2 | 15 | 2 | 16 | 21 | 41 | 12 | 19 | 40
Anxiety (Psychiatric disorders) | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 4 | 3 | 1 | 6 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4 | 0 | 7 | 0 | 6 | 9 | 26 | 8 | 13 | 24
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 2 | 3 | 1 | 2 | 8 | 13 | 0 | 10 | 12
Acne (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0 | 2 | 1 | 0 | 5 | 7 | 2 | 6 | 9
Rash (Skin and subcutaneous tissue disorders) | 5 | 2 | 4 | 1 | 7 | 2 | 5 | 5 | 22 | 5 | 12 | 20
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 2 | 2 | 2 | 3 | 0 | 1 | 2

LIMITATIONS AND CAVEATS:
The global study was interrupted due to issues with the clinical supply.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.